CLINICAL TRIAL: NCT01466478
Title: A Phase I Exploratory Study Evaluating 3 Formulations of LEO 29102 Plus Calcipotriol, Ointment, LEO 29102 Ointment, Calcipotriol Ointment, Daivonex® Ointment and Diprosone® Ointment in the Treatment of Psoriasis
Brief Title: An Exploratory Psoriasis Plaque Test Study With LEO 29102 Plus Calcipotriol, Ointment, in Psoriasis Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: PLQ-007; 2011-003058-25
Record Dates: First submitted 2011-10-26; First posted 2011-11-08 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2013-10

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene; Ointments

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- LEO 29102 plus calcipotriol (Experimental)
  Interventions: Drug: Ointment A: LEO 29102 2.5 mg/g plus calcipotriol 50 µg/g ointment; Drug: Ointment B: LEO 29102 2.5 mg/g ointment; Drug: Ointment C: Calcipotriol 50 µg/g ointment; Drug: Ointment D: LEO 29102 2.5 mg/g plus calcipotriol 50 µg/g ointment; Drug: Ointment G: LEO 29102 2.5 mg/g plus calcipotriol 50 µg/g ointment; Drug: Daivonex® ointment; Drug: Diprosone® ointment

INTERVENTIONS:
Drug: Ointment A: LEO 29102 2.5 mg/g plus calcipotriol 50 µg/g ointment — once daily application, 4 weeks
Drug: Ointment B: LEO 29102 2.5 mg/g ointment — once daily application, 4 weeks
Drug: Ointment C: Calcipotriol 50 µg/g ointment — once daily application, 4 weeks
Drug: Ointment D: LEO 29102 2.5 mg/g plus calcipotriol 50 µg/g ointment — once daily application, 4 weeks
Drug: Ointment G: LEO 29102 2.5 mg/g plus calcipotriol 50 µg/g ointment — once daily application, 4 weeks
Drug: Daivonex® ointment — once daily application, 4 weeks
Drug: Diprosone® ointment — once daily application, 4 weeks

SUMMARY:
The purpose of the study is to compare the 3 ointment formulations containing LEO 29102 plus calcipotriol and Daivonex® ointment and Diprosone® ointment and to compare LEO 29102 plus calcipotriol to LEO 29102 alone and to calcipotriol alone in the same ointment vehicle, using the psoriasis plaque test modified from the method developed by KJ Dumas and JR Scholtz.

ELIGIBILITY:
Inclusion Criteria:

* Following verbal and written information about the trial, the subject has to provide signed and dated informed consent before any study related activities are carried out.
* Age 18 years or above.
* Either sex.
* All skin types.
* Outpatients with a diagnosis of psoriasis vulgaris with lesions located on arms, legs and/or trunk. The lesions must have a total size suitable for application of 7 different products.
* Subjects with, in the opinion of the investigator, stable psoriasis based on Total Plaque Score evaluated at screening visit and at visit 2 (Baseline).
* Subjects with psoriasis lesions (plaques) assessed by a Total Clinical Score (sum of scores of erythema, scaling and infiltration) of 4 to 9 inclusive but each individual item ≥ 1.
* Subjects willing and able to follow all the study procedures and complete the whole study.
* Subjects affiliated to a social security system.
* Female subjects of childbearing potential using a reliable method of contraception for at least 1 month before the study start and during the course of the study (e.g., oral contraceptive pill, intrauterine device, contraceptive patches, implantable contraception, condoms) or females of non childbearing potential (i.e. postmenopausal (absence of menstrual bleeding for 2 years), hysterectomy, bilateral ovariectomy or tubal section/ligation).
* Female with a negative urine pregnancy test at Visit 1 (screening visit).

Exclusion Criteria:

* Females who are pregnant, of child-bearing potential and who wish to become pregnant during the study, or who are breast feeding.
* Systemic treatment with biological therapies (marketed or not marketed) with a possible effect on psoriasis vulgaris within 4 weeks (etanercept), 2 months (adalimumab, alefacept, infliximab), 4 months (ustekinumab) or 4 weeks/5 half-lives (which-ever is longer) for experimental biological products prior to randomisation and during the study.
* Systemic treatments with all other therapies than biologicals, with a potential effect on psoriasis vulgaris (e.g., corticosteroids, retinoids, immunosuppressants) within the 4-week period prior to randomisation and during the study.
* Use of phototherapy within the following time periods prior to randomisation and during the study:

  * PUVA (4 weeks),
  * UVB (2 weeks).
* Subjects using one of the following topical drugs for the treatment of psoriasis within the 4 week period prior to randomisation and during the study:

  * Potent or very potent (WHO group III-IV) corticosteroids.
* Subjects using one of the following topical drugs for the treatment of psoriasis within two weeks prior to randomisation and during the study:

  * WHO group I-II corticosteroids (except if used for treatment of scalp and/or facial psoriasis),
  * Topical retinoids,
  * Vitamin D analogues,
  * Topical immunomodulators (e.g. macrolides),
  * Anthracen derivatives,
  * Tar,
  * Salicylic acid.
* Subjects using emollients on the target plaques within one week before randomisation and during the study.
* Initiation of, or expected changes to concomitant medication that may affect psoriasis vulgaris (e.g., beta blockers, anti-malaria drugs, lithium and ACE inhibitors) within 2 weeks prior to the randomisation and during the study.
* Subjects with current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis.
* Subjects with known/suspected disorders of calcium metabolism associated with hypercalcemia within the last 10 years, based on medical history and/or subject interview.
* Subjects with any of the following conditions present on the test area: viral (e.g. herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections and atrophic skin.
* Subjects with skin manifestations in relation to syphilis or tuberculosis, rosacea, perioral dermatitis, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, acne rosacea, ulcers and wounds within the plaque test areas.
* History of any severe disease or serious current condition (based on subject interview and/or results of screening physical examination) which, in the opinion of the Investigator, would put the subject at risk by participating in the study or would interfere significantly with the evaluation of study results or the study course (e.g. cancer, severe cardiopathy, severe renal insufficiency, severe hepatic insufficiency).
* Subjects who have received treatment with any non-marketed drug substance (i.e., an agent which has not yet been made available for clinical use following registration) within the 4 week period prior to randomisation or longer, if the class of the substance requires a longer washout as defined above (e.g., biological treatments).
* Subjects with current participation in any other interventional clinical trial, based on interview of the subject.
* Subjects with known or suspected hypersensitivity to component(s) of the investigational product(s).
* Subjects with any concomitant medical or dermatological disorder(s) which might preclude accurate evaluation of the psoriasis on the test areas.
* Subjects foreseeing an intensive solar exposure during the study (UV radiation, etc.) or having been exposed within two weeks preceding the screening visit.
* Subjects impossible to contact in case of emergency.
* Subjects who are known or, in the opinion of the investigator, are unlikely to comply with the Clinical Study Protocol (e.g. alcoholism, drug dependency or psychotic state).
* Subjects who are in an exclusion period in the National Biomedical Research Register of the French Ministry of Health at randomisation.
* Subjects under guardianship, hospitalized in a public or private institution, for a reason other than the research or subject deprived of freedom.
* Subjects previously randomised in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of treatment in Total Clinical Score (TCS) of clinical symptoms (sum of erythema, scaling and infiltration). | 4 weeks
  TCS range from 0 (all symptoms absent) to 9 (all symptoms severe)

SECONDARY OUTCOMES:
Clinical criteria: - Change from baseline in single clinical symptom score: erythema, scaling, infiltration at end of treatment and individual visits, - Change from baseline in Total Clinical Score (TCS) at individual visits. | 4 weeks
Ultrasonography: Change from baseline to end of treatment in lesion thickness (total and echo-poor band) measured by ultrasound. | 4 weeks
NIR spectroscopy: Change from baseline to Day 15 and end of treatment in the ratio between the peaks at 6900 cm-1 and at 5200 cm-1, the width of the peak at 6900 cm-1 and the calculated severity score | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Queille-Roussel, MD, Principal Investigator — Centre de Pharmacologie Clinique Appliquée à la Dermatologie (CPCAD)
Locations (1):
- CPCAD - Centre de Pharmacologie Clinique Appliquée à la Dermatologie, Nice, France

IPD SHARING:
Plan to Share IPD: No